CLINICAL TRIAL: NCT05616715
Title: Evaluation of Different Periodontal Plastic Surgery Techniques for Gummy Smile Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHDFPS
Record Dates: First submitted 2022-09-22; First posted 2022-11-15 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-09

CONDITIONS: Gummy Smile
MeSH Terms: interventions — Crown Lengthening; Gingivectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects with gummy smile and with upper lip hypermobility (Experimental): Periodontal plastic surgery for peek device implantation with 4 screws in the anterior maxillary area
  Interventions: Device: Peek device
- Subjects with gummy smile and with short teeth and upper lip hypermobility (Experimental): Gingivectomy/crown lengthening and device implantation in the anterior maxillary area. First crown lengthening procedure (CLP) will be performed creating a distance of 3mm between cementoenamel junction (CEJ). Next peek device will be position with 4 screws
  Interventions: Device: Peek device
- Patiens who refuse device implantation - control group (Experimental): Gingivectomy/crown lengthening procedure
  Interventions: Other: Crown lengthening/gingivectomy

INTERVENTIONS:
Device: Peek device — Participants with gummy smile will be recruited from the Dental Clinic of Instituto Universitário Egas Moniz
  Arms: Subjects with gummy smile and with short teeth and upper lip hypermobility; Subjects with gummy smile and with upper lip hypermobility
Other: Crown lengthening/gingivectomy — Participante with gummy smile will be recruited from the Dental Clinic of Instituto Universitário Egas Moniz
  Arms: Patiens who refuse device implantation - control group

SUMMARY:
Investigating different periodontal surgery techniques to treat gummy smile.

DETAILED DESCRIPTION:
Participants will be subdivided into 3 (three) groups:

1. Patients with upper lip hypermobility - surgery for device implantation in the anterior area of the maxilla;
2. Patients with short teeth and upper lip hypermobility - flap surgery/gingivectomy and device implantation; and
3. Patients who refuse implantation - flap surgery/gingivectomy;

ELIGIBILITY:
Inclusion Criteria:

* Gummy smile due to two etiologies (combined or isolated);
* Short clinical crown of teeth due to the altered passive eruption;
* Upper lip hyperactivity

Exclusion Criteria:

* Smokers;
* Pregnant or breastfeeding patients;
* Patients with systemic diseases that can affect the result of surgical treatment (such as diabetes, heart diseases and taking blood anticoagulant medication, blood diseases, immunodeficiency disease etc.);
* Cleft lip;
* Craniofacial syndrome;
* Facial alteration surgeries during the study;
* Active orto treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Superior incisors proportion (height x length) | Baseline and week 24
  Superior incisors height and lenght
Change in Exposure of central incisors at rest | Baseline and week 24
  Measurement between incisal border of central incisors and the border of the lower lip during smile (in millimeters)
Change in Periodontal probing | Baseline and week 24
  Three probes (mesial, buccal and distal) for exposed teeth during smile
Change in Gengiva exposure at rest and forced smile | Baseline and week 24
  When lips are in rest position measure the amount of exposed gingiva and during a forced smile, make the same measure
Change in Interlabial space at rest | Baseline and week 24
  When in rest position, measure distance between lips

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz Cooperativa de Ensino Superior, Almada, Portugal

IPD SHARING:
Plan to Share IPD: No